CLINICAL TRIAL: NCT03653273
Title: Disease Modifying Therapies Withdrawal in Inactive Secondary Progressive Multiple Sclerosis Patients Older Than 50 Years
Brief Title: Disease Modifying Therapies Withdrawal in Inactive Secondary Progressive Multiple Sclerosis Patients Older Than 50 Years (STOP-I-SEP)
Acronym: STOP-I-SEP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC17_8842_STOP-I-SEP
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; secondary progressive; disease modifying treatment; medico economic impact; treatment withdrawal
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DMT withdrawal (Experimental): DMT will be immediately stopped after randomization.These patients will be followed for 2 years.
  Interventions: Other: DMT withdrawal
- DMT continuation (Active Comparator): The previously established therapy will be continued at the same dose during two years.
  Interventions: Drug: DMT continuation

INTERVENTIONS:
Other: DMT withdrawal — Group 1 (DMT withdrawal) will not undergo any disease modifying treatments (DMT).
  Arms: DMT withdrawal
Drug: DMT continuation — Group 2 (DMT continuation) may undergo the DMT . The therapy continued in this research is the one previously established, at the same dose, not implying additional precautions for use.
  Arms: DMT continuation

SUMMARY:
Further controlled and randomized prospective studies in Multiple sclerosis, analyzing the potential impact of treatment discontinuation on disability progression, focal disease activity and quality of life are needed. The optimum patient age and duration of inactive SPMS before treatment withdrawal and the monitoring procedures also need to be specified, the ultimate goal being to provide evidence-based recommendations for clinical practice. Following the previous retrospective experience, we decided to drive a multicenter prospective study in France based on the hypothesis that stopping disease modifying therapy will not induce an increased risk of disability progression and relapse in selected SPMS patients (older patients without lesion activity) but will improve the quality of life and may reduce treatment-related costs.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) usually evolves over decades and can present several phenotypes. Approximately 85% of newly diagnosed Multiple Sclerosis (MS) patients present the Relapsing-Remitting MS (RRMS) phenotype. After a mean time of approximatively 20 years, a large majority of these patients evolve to the so-called "Secondary Progressive MS" (SPMS) phase. SPMS is characterized by an irreversible disability progression not related to relapses, although relapses could be superimposed. Nevertheless, the shift in-between RRMS and SPMS is not clear. Different subtypes of SPMS have been recently defined by F Lublin et al. This classification takes into account persistent focal inflammatory activity (active vs inactive SPMS) along with disease progression (progressing vs non-progressing SPMS). In clinical routine, it is important to identify these stages of MS as they differently respond to the disease modifying therapies (DMTs).

Introducing DMTs during the RRMS phase had consistently demonstrated a significant impact on the annual relapse rate (ARR) and on the short-term disability progression. Conversely, during the SPMS phase, the impact of DMTs remained uncertain on disability progression, especially in older patients, with "inactive" disease. As a matter of fact, the DMTs are considered to be anti-inflammatory by nature, but the focal inflammation reduces with age and disease duration.

In addition, the DMTs have side effects and cost approximately 10,000 euros per year and per patient. In this context, the usefulness of continuing DMTs in "inactive" SPMS patients older than 50 years is questionable.

In a preliminary retrospective study conducted at our Institute which enrolled 100 SPMS patients, the ARR remained stable 3 years after treatment withdrawal (0.07, 95% CI [0.05, 0.11]), relative to the 3 years prior to treatment withdrawal (0.12, [0.09, 0.16]). EDSS scores were available for 94 patients The percentage of patients experiencing a significant increase of their EDSS score during the 3 years after treatment withdrawal also remained stable compared to the 3 years prior treatment withdrawal. These preliminary data support the safety of DMTs withdrawal in selected SPMS patients. However, further prospective studies are needed to provide evidence-based guidelines for daily practice.

This randomized controlled clinical trial thus aims to compare SPMS patients older than 50 years without evidence of focal inflammatory activity for 3 years, stopping DMTs versus patients with the same criteria still receiving treatment. We hypothesize that stopping DMTs will not induce an increased risk of disability progression or relapse in SPMS patients but will improve their quality of life and have an impact on treatment-related costs.

So far, the impact of DMTs withdrawal in a selected SPMS population has not been explored. Having evidence-based recommendations on the treatment management of these patients is essential, considering the consequences in terms of disability, relapses, side effects, quality of life and costs. DMTs in MS are now available since 20 years, with an increasing number of approved molecules. As a matter of fact, this question concerns a large number of patients: a retrospective analysis of patients included in the Rennes EDMUS database allowed to identify 71 SPMS patients older than 50 years and without evidence of focal inflammatory activity for 3 years actually undergoing a DMT.

For evident conflict of interests, the pharmaceutical firms will not promote or fund clinical trials on treatment withdrawal. A randomized controlled study initiated by academia and financed by public funding should be performed to explore these questions. We will evaluate the impact of these changes from the patient and the health system's points of view. The results of this clinical trial will lead to a concrete change in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 50 years old;
* Secondary progressive phenotype for at least 3 years; The secondary progressive phenotype will be defined as progressive deterioration of disability not due to relapse, with an increase of at least 1 EDSS point since the beginning of the progressive phase (or 0.5 EDSS point if EDSS score ≥ 5.5).
* Disease modifying therapy of MS for at least 3 years (interferon, glatiramer acetate, teriflunomide, dimethyl fumarate, cyclophosphamide, azathioprine, methotrexate, mycophenolate mofetil, rituximab, ocrelizumab); Both patients with the same DMT or with successive DMTs during 3 years can be included. It is important to note that patients could have been treated with fingolimod or natalizumab 2 or 3 years before inclusion, but not during the year before inclusion ;
* No evidence of focal inflammatory activity for at least 3 years (no clinical relapse and no gadolinium enhancement on an MRI scan);
* EDSS≥3.

Concomitant medications with Fampridine are allowed throughout the study, provided they have been introduced at least 1 months before inclusion.

Natalizumab and fingolimod during the year before inclusion were excluded because of the risk of recurrence of inflammatory activity or even rebound of inflammatory activity after withdrawal.

Both patients with the same DMT or with successive DMTs during 3 years can be included, as for example, cyclophosphamide is used for 1 or 2 years, sometimes followed by mycophenolate mofetil.

For Rituximab and Ocrelizumab, inclusion in STOP-I-SEP will be at 6 months from the last infusion to take into account the mode of action of these treatments and their specific administration scheme.

Exclusion Criteria:

* Patients treated with mitoxantrone or alemtuzumab, during the previous 3 years before inclusion;
* Patients treated with natalizumab or fingolimod during the year before inclusion;
* Change of disease modifying therapy of MS for less than a year
* Other neurological or systemic disease ;
* Incapacity to understand or sign the consent form ;
* Contraindication to MRI ;
* Pregnancy or breast-feeding ;
* Patient in another clinical trial
* Persons referred to in Articles L. 1121-5 to L. 1121-8 and L. 1122-1-2 of the Public Health Code (eg minors, protected adults, …).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Disability progression measured by EDSS | 24 months
  Disability progression measured by the Percentage of patients experiencing disability progression (confirmed at 6 months) at 2 years.
  Disability progression will be defined as an increase in the EDSS of at least 1 point if the baseline EDSS was 5.5 or less, or 0.5 point if the Baseline EDSS was more than 5.5.

SECONDARY OUTCOMES:
Time of Disability progression | 24 months
  Disability progression measured by Time from DMT withdrawal to disability progression
Disability progression measured by composite score | 24 months
  Disability progression measured by Change in a composite disability progression score (increase in the EDSS score, or an increase in the time to perform the timed 25-foot walk ≥ 20%, or an increase in the time to complete the 9-hole peg test ≥ 20%) confirmed at 6 months
Disability progression measured by SDMT | 24 months
  Disability progression measured by Change in the SDMT score from baseline to 2-year
Percentage of patients with Relapse | 24 months
  Relapses measured by Percentage of patients with at least one relapse from baseline to 2-year
Annualized relapse rate | 24 months
  Relapses measured by Annualized relapse rate during 2-year
Time of Relapses | 24 months
  Relapses measured byTime from DMT withdrawal to first relapse;
Percentage of patients with brain lesion | 24 months
  Percentage of patients with one or more new or enlarging brain MRI (Magnetic Resonance Imaging) lesions from baseline to 2-year
Percentage of patients with gadolinium enhancing lesion | 24 months
  Percentage of patients with at least one gadolinium enhancing lesion(s) at 6 months, and/or 1 year,and/or 2-year
Change in brain volume | 24 months
  Change in brain volume from baseline to 2-year measured on MRI
Percentage of patients with no evidence of disease activity | 24 months
  Percentage of patients with no evidence of disease activity (NEDA 3: no clinical relapse, no MRI activity, no disability progression) at 2-year
Percentage of patients who resume DMT in the treatment withdrawal group | 24 months
  Percentage of patients who resume DMT in the treatment withdrawal group at 2-year
Quality of life measured by SEP-59 score | 24 months
  Change in the SEP-59 score from baseline to 2-year;
Quality of life measured by EQ-5D score | 24 months
  Change in the EuroQOL EQ-5D from baseline to 2-year;
Medico economic impact | 24 months
  Incremental Cost Effectiveness Ratio (ICER) defined as the cost for QALY gained in "treatment withdrawal group" versus "treatment continued group"

CONTACTS AND LOCATIONS:
Overall Officials: Anne KERBRAT, Dr, Principal Investigator — CHU Rennes - National Headache Center; Clarisse SCHERER-GAGOU, Dr, Principal Investigator — University Hospital, Angers; Jean PELLETIER, Pr, Principal Investigator — AP-HM; Céline LOUAPRE, Dr, Principal Investigator — AP-HP La pitié Salpêtrière; Aurore JOURDAIN, Dr, Principal Investigator — CHU Brest; Pierre CLAVELOU, Pr, Principal Investigator — University Hospital, Clermont-Ferrand; Thibault MOREAU, Pr, Principal Investigator — CHU Dijon; Olivier CASEZ, Dr, Principal Investigator — University Hospital, Grenoble; Hélène ZEPHIR, Pr, Principal Investigator — CHU Lille; Sandra VUKUSIC, Pr, Principal Investigator — Hospices Civils de Lyon; Pierre LABAUGE, Pr, Principal Investigator — University Hospital, Montpellier; Guillaume MATHEY, Dr, Principal Investigator — CHU NANCY; David LAPLAUD, Pr, Principal Investigator — Nantes University Hospital; Christine LEBRUN-FRENAY, Pr, Principal Investigator — CHU NICE; Olivier HEINZLEF, Dr, Principal Investigator — CH Poissy; Jean-Philippe NEAU, Pr, Principal Investigator — CHU Poitiers; Marc COUSTANS, Dr, Principal Investigator — CH Quimper; Jérôme DE SEZE, Pr, Principal Investigator — CHU Strasbourg; Anne-Marie GUENNOC, Dr, Principal Investigator — CHU Tours; Caroline BENSA-KOSCHER, Dr, Principal Investigator — Fondation de Rothschild; Eric THOUVENOT, Pr, Principal Investigator — Centre Hospitalier Universitaire de Nīmes; Alain CREANGE, Pr, Principal Investigator — CH HENRI MONDOR; Arnaud KWIATKOWSKI, Dr, Principal Investigator — Hôpital Saint Vincent de Paul; Aurelie RUET, Pr, Principal Investigator — University Hospital, Bordeaux; Jérôme GRIMAUD, Dr, Principal Investigator — CH de Chartres; Maia TCHIKVILADZE, Dr, Principal Investigator — CH Foch; Philippe CASENAVE, Dr, Principal Investigator — CH de Libourne
Locations (27):
- France (27):
  - CHU Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CH de Chartres, Chartres
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CH de Libourne, Libourne
  - CHU Lille, Lille
  - Hôpital Saint Vincent de Paul, Lille
  - Hospices Civils Lyon, Lyon
  - AP-HM, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU de Nîmes, Nîmes
  - AP-HP (La Pitié Salpêtrière), Paris
  - Fondation de Rothschild, Paris
  - CH Poissy, Poissy
  - CHU Poitiers, Poitiers
  - CH Quimper, Quimper
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - CH de Foch, Suresnes
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No